CLINICAL TRIAL: NCT06228651
Title: The Functional Outcome of the Arterial Tourniquet in Total Knee Arthroplasty- a RCT of Bilateral Total Knee Arthroplasties.
Brief Title: The Effect of the Tourniquet in Bilateral Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: s-20150100
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Tourniquet and Outcome After Total Knee Replacement
Keywords: Tourniquet, Total knee replacement, Oxford knee score, Forgotten Joint Score
MeSH Terms: interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: We conducted a prospective, randomized, double -blinded trial including patients with simultaneously performed bilateral TKA in a fast-track setup at Lillebaelt Hospital - Vejle, Denmark. After randomization, tourniquet was inflated to only one knee facilitating direct comparison with patients acting as their own controls. Postoperative evaluations were performed at predetermined intervals. Patient reported outcomes were measured for the following year postoperative
Who Masked: Participant, Investigator
Masking Description: The protocol for tourniquet application during TKA began with encasing the patient's thigh in a stockinette sleeve, followed by the fitting of the tourniquet cuff which was connected to the Zimmer A.T.S 3000 tourniquet system. To ascertain the individualized optimal pressure, a pulse oximeter was momentarily placed on the patient's limb before the cuff was inflated. The tourniquet was used from the start of the incision and was released just prior to closure of the joint capsule to ensure optimal hemostasis during the final stages of the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tourniquet (Active Comparator): The leg with the tourniquet which was inflated during surgery
  Interventions: Device: Tourniquet
- Control (Active Comparator): The leg without the tourniquet which was not inflated during surgery
  Interventions: Other: The leg without the tourniquet

INTERVENTIONS:
Device: Tourniquet
  Arms: Tourniquet
Other: The leg without the tourniquet
  Arms: Control

SUMMARY:
This study describes in a randomised controlled trial how the tourniquet influence the outcome af a total knee replacements

DETAILED DESCRIPTION:
Background: Tourniquet application during total knee arthroplasty (TKA) is a common practice aimed at reducing intraoperative bleeding. However, concerns have been raised about potential tissue damage from ischemia and reperfusion injury.

Objectives: This study examines the effects of tourniquet use during TKA on postoperative functional outcomes, including pain, range of motion (ROM), and patient-reported outcomes (PROMs).

Methods: In a fast-track surgical setting, a prospective, randomized, double-blinded trial was conducted with patients undergoing bilateral TKA. Tourniquets were applied to one knee, while the contralateral knee served as a control. Evaluations were conducted at two and four weeks, and at three and twelve months postoperatively, employing paired t-tests and mixed-effects linear modeling for data analysis.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 years or older, planned for bilateral cemented primary TKA due to osteoarthritis during the same session. and showed a uniform degree of osteoarthritis determined by the Kellgren-Lawrence classification

Exclusion Criteria:

non-Danish speaking patients, unable to cooperate for VAS scoring, coagulation disorders, salicylate-induced asthma, severe thrombocytopenia, serious heart failure, severe liver failure, hypovolemia (any cause), dehydration, angioedema, bronchospasm, undergoing lithium treatment, suspected or manifest gastrointestinal bleeding, cerebrovascular bleeding, high postoperative bleeding risk or delayed hemostasis, hypersensitivity to adrenaline, sympathomimetics or excipients , hypertrophic or ischemic heart disease, undergoing dihydroergotamine treatment and thyrotoxicosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 2 weeks postoperatively
  Pain at rest evaluated at a visual analogue scale (VAS)

SECONDARY OUTCOMES:
Forgotten Joint Score (FJS) and Oxford Knee Score (OKS) | two weeks, four weeks, three months and one year postop
  Patient reported outcome
Wound complications and deep vein thrombosis and re-admissions | within one year postop

IPD SHARING:
Plan to Share IPD: No